CLINICAL TRIAL: NCT01583595
Title: Determining the Relationships Between Self-efficacy for Walking Ability, Gate Speed and Physical Activity in Patients With Chronic Lung Disease
Brief Title: Self Efficacy, Walking Ability, Gait Speed and Physical Activity in People With Chronic Lung Disease
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Roberto P. Benzo, Consultant Pulmonary and Critical Care Medicine, Mayo Clinic
Other Study IDs: 11-008157
Record Dates: First submitted 2012-02-07; First posted 2012-04-24 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Lung Disease; Self-efficacy
Keywords: Chronic Lung Disease; Exercise; Self-efficacy
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Most patients with chronic lung disease underestimate their actual walking ability due to low confidence. To better understand the relationships between lung function, self-efficacy for walking (confidence in ability to walk a defined distance), actual walking ability for the same distance gait speed and physical activity level-PAL- (total energy expenditure/resting metabolic rate).

Quality of life, self efficacy for activity questionnaires, physical activity level measurement, 4-meter gait speed and 6-minute walk distance will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 40 years and older
* Diagnosis of any chronic lung disease as evidenced by pulmonary function testing completed within the prior 12 months
* Able to walk independently and successfully complete the 6-minute walk assessment

Exclusion Criteria:

* Unable to walk without assistance or complete the 6-minute walk assessment
* Patients unable to comprehend and accurately respond to the study questionnaires either by written or spoken communication
* Patients diagnosed with or treated for a lower respiratory tract infection or COPD exacerbation within the prior 30 days

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic lung disease
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Analyze associations between self-efficacy for walking, gait speed, physical activity level and perceptions of symptoms in patient with chronic lung disease (COPD and Pulmonary Fibrosis) | Day of enrollment.
  Correlation , regression models and mediation analysis (self efficacy and physical activity) will be performed.

SECONDARY OUTCOMES:
Predictive utility of 4-meter gait speed for estimating physical activity level (PAL) as validated by gold standard activity monitor. | 1 week
  Measure 4-meter gait speed during standardized 6 mintute walk test and compare to armband activity monitor results to determine predictive ability, if any, on PAL in people with chronic lung disease.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto P Benzo, M.D., MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States